CLINICAL TRIAL: NCT02020382
Title: Evaluation of the Diagnostic Value of microRNAs for Inflammatory Bowel Disease
Brief Title: Evaluation of the Diagnostic Value of microRNAs for Inflammatory Bowel Diseases
Acronym: MicroMICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P120903; 2013-A00310-45 (Other: IDRCB)
Record Dates: First submitted 2013-12-09; First posted 2013-12-24 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Ulcerative Colitis; Crohn Disease; Healthy; Non-IBD Colitis
Keywords: microRNAs; IBD; Crohn's disease; Ulcerative colitis; colonic polyps screening; controls
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Crohn adult colic (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS
- RCH adults (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS
- Witnesses healthy adults (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS
- Witnesses adults with non-IBD inflammation (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS
- Children with colitis (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS
- Witnesses healthy children (Other): testing qPCR diagnostic KIT of microRNAS from colonic biopsies
  Interventions: Device: qPCR diagnostic KIT of microRNAS

INTERVENTIONS:
Device: qPCR diagnostic KIT of microRNAS — testing qPCR diagnostic KIT of microRNAS from colonic biopsies

SUMMARY:
The purpose of this study is to assess the diagnostic value of microRNAs in IBD colon (ulcerative colitis or Crohn's disease) in adults as compared to healthy controls (and non-IBD colitis)

DETAILED DESCRIPTION:
RATIONAL Inflammatory Bowel Disease (IBD) affects more than 200,000 people in France and 1.5 million in Europe. Difficulties in the management of IBD are related to the need for invasive tests for the diagnosis of IBD (endoscopy), partly explaining the delay in diagnosis, and the inability to distinguish early colonic Crohn's disease of ulcerative colitis (UC) in 10-30% of cases.

Recently, we identified real-time polymerase chain reaction (PCR), from healthy colonic mucosa of IBD patients, a molecular signature of IBD involving 10 microRNA (miRNA) Common (miR26a, miR29a, miR29b, miR126 * miR15a, miR127-3p, miR324 -3p, miR30c, miR185, miR196a) and 15 colic chronic disease (MC) and ulcerative colitis (RCH) discriminating microRNA (miR-142-3p, miR-142-5p, miR-146a, miR-146b-5p, miR150, miR-181d, miR-182, miR199a -3p, miR199a-5p, miR199b-5p, miR-203, miR223, miR-299-5p, miR320a, miR-328).

TYPE OF STUDY : multicenter diagnostic evaluation Study

MAIN PURPOSE OF THE STUDY : To evaluate the diagnostic value of microRNA in colonic IBD (ulcerative colitis or Crohn's disease) in adults as compared to healthy controls (and non-IBD colitis)

SECONDARY OBJECTIVES :

* assess the ability of microRNA to discriminate a colic chronic disease (MC) of ulcerative colitis (RCH) in adults
* evaluate the diagnostic value of microRNA in inflammatory colitis child
* explore the possibility of measuring miRNA of interest in the stool

PRODUCTS OF THE STUDY diagnostic kit of IBD in quantitative polymerase chain reaction (qPCR)

NUMBER OF PATIENTS : 6 groups of 50 patients each will be included

* Group 1: Crohn adult colic
* Group 2: ulcerative colitis (RCH) adults
* Group 3: Witnesses healthy adults
* Group 4: Witnesses adults with non-IBD inflammation
* Group 5: Children with colitis
* Group 6 : Witnesses healthy children

INCLUSION LENGTH 30 months

DURATION OF THE STUDY 30 months

ELIGIBILITY:
Inclusion criteria :

* Target Population : Patients (children and adults), man or woman, suffering from Crohn's disease with colonic involvement or ulcerative colitis according to the criteria of the European consensus (ECCO 2010)
* Control population: healthy subjects and any non-Crohn's colitis or ulcerative colitis
* Having a colonoscopy examination indication,
* Who signed the consent form (for adults and signed parental consent obtained for patients minors)

Exclusion Criteria:

* No health insurance ,
* mental disability,
* pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic value of microRNAs in qPCR,in IBD colon (ulcerative colitis or Crohn's disease) in adults compared to health | 1 day
  Evaluate the diagnostic value of microRNAs in qPCR, suitable for routine use, initially testing the expression of 25 miRNAs from endoscopic biopsies in IBD colon (ulcerative colitis or Crohn's disease) in adults compared to health

SECONDARY OUTCOMES:
- Evaluate the ability of miRNAs to discriminate a MC colic of UC in adults | 1 day
Evaluate the diagnostic value of microRNAs in inflammatory colitis child | 1 day
- Study the possibility of measuring miRNA of interest in feces and saliva | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Treton, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (5):
- France (5):
  - Hôpital Beaujon, Clichy
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Robert Deré, Paris

IPD SHARING:
Plan to Share IPD: Undecided